CLINICAL TRIAL: NCT06186310
Title: Effectiveness of Aquatic Therapy on Balance and Functionality in Children With Duchenne and Becker Muscular Dystrophy
Brief Title: Effectiveness of Aquatic Therapy in Children With Duchenne and Becker Muscular Dystrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Ceyda Ulu, Assistant doctor in the department of physical medicine and rehabilitation, Gaziosmanpasa Research and Education Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GaziosmanpasaTREH-FTR-CU-01
Record Dates: First submitted 2023-12-15; First posted 2024-01-02 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Duchenne or Becker Muscular Dystrophy
Keywords: Aquatic Exercise Therapy; Muscular Dystrophy; Life Quality; Functional Status; Balance Control
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies

STUDY DESIGN:
Intervention Model Description: Two groups with a conventional physical therapy control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aquatic Therapy Group (Active Comparator): in addition to the home programme exercises, aquatic exercises will be performed with a physiotherapist
  Interventions: Other: Aquatic Therapy Group
- Conventional Physical Therapy Group (Active Comparator): Personalized exercises in the form of a home program will be demonstrated by the physiotherapist
  Interventions: Other: Conventional Physical Therapy Group

INTERVENTIONS:
Other: Aquatic Therapy Group — After the initial evaluations, patients will be given aquatic exercises including personalized strengthening, balance and breathing exercises accompanied by a physiotherapist 3 days a week for total 5 weeks. At the same time, the exercises taught as a home program will be asked to be repeated every day for 5 weeks.
  Arms: Aquatic Therapy Group
Other: Conventional Physical Therapy Group — After the initial evaluations, patients in the control group will be taught passive, active, actively assisted or resistant upper and lower extremity exercises as a home program, appropriate to each patient's functional level and muscle strength. Subjects will be asked to perform the exercises every day for 5 weeks, not exceeding an average of 45 minutes, 5 to 10 repetitions of each exercise, depending on fatigue.
  Arms: Conventional Physical Therapy Group

SUMMARY:
The purpose of this study is ; to evaluate the effects of aquatic therapy applied in addition to conventional physical therapy on balance, functionality and quality of life in children with Duchenne and Becker muscular dystrophy.

DETAILED DESCRIPTION:
Duchenne and Becker muscular dystrophy is the most common type of muscular dystrophy in childhood caused by a mutation of the DMD gene. Progressive muscle weakness is the main symptom, as muscle fiber degeneration is the primary pathological process.

Weakness selectively affects the proximal before the distal limb muscles and the lower before the upper limbs. The affected child therefore has difficulty running, jumping, and walking up steps.

Although there is currently no treatment method that eliminates the disease, exercise practices significantly improve the quality of life of children.

There are not enough studies in the literature evaluating whether the addition of aquatic therapy to conventional physical therapy helps to improve balance skills, functionality and quality of life in children with muscular dystrophy.

The purpose of this study is ; to evaluate the effects of aquatic therapy applied in addition to conventional physical therapy on balance, functionality and quality of life in children with Duchenne and Becker muscular dystrophy.

Our study will include children aged 5-18 years and complete a 10 -m walk without assistance/support who are diagnosed with Duchenne or Becker muscular dystrophy by a neurologist and followed up in the Muscular Diseases Unit of Gaziosmanpaşa Training and Research Hospital In follow-ups, patients who are planned to receive aquatic therapy will be listed according to their application dates.

In addition to the exercises home programme, patients at the top of the list will receive aquatic treatment 3 days a week for a total of 5 weeks with a physiotherapist.

Patients at the bottom of the list will form the control group and will receive home programme exercise while waiting in line for aquatic therapy After 5 weeks, the initial assessments will be repeated and recorded

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Duchenne Muscular Dystrophy or Becker Muscular Dystrophy by a neurologist
* Between the ages of 5-18, with ongoing ambulation
* Co-operating with the physiotherapist's practices

Exclusion Criteria:

* Those who will not be able to perform the evaluation parameters
* Have a serious systemic disease that may interfere with exercise
* Injury and/or surgery in the last 6 months
* Receive gene therapy
* In the presence of contraindications to aquatic therapy such as excessive fear of water, behavioral problems, shortness of breath at rest, infection, incontinence, known chlorine allergy, open wound, acute systemic disease, epilepsy, tracheotomy, permanent drain, immunodeficiency

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2023-11-05 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Pediatric Berg Balance Scale | five weeks
  The Pediatric Balance Scale is a modified version of the Berg Balance Scale that is used to assess functional balance skills in school-aged children. The scale consists of 14 items: sitting to standing,standing to sitting,transfers,standing unsupported,sitting unsupported,standing with eyes closed,standing with feet together,standing with one foot in front,standing on one foot,turning 360 degrees,turning to look behind,retrieving object from floor,placing alternate foot on stool,reaching forward with outstretched arm. That are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points.

SECONDARY OUTCOMES:
Timed Performance Tests (walking 10 m, climbing 4 steps and descending 4 steps) | five weeks
  It will be used to evaluate the functional performance of children against time.
  Time to climb a 4-step staircase: They will be asked to climb a 4-step stair platform in the same way they climb in daily life
  Descending a 4-step ladder: They will be asked to descend a 4-step ladder platform in the same way they descend in daily life.
  Time to walk a distance of 10 meters: Children are asked to walk a predetermined distance of 10 meters at the same pace they walk in their daily lives.Results will be recorded.
The Pediatric Quality of Life Inventory (PedsQL)-Neuromuscular Module (PedsQL-3.0 | five weeks
  The PedsQL 3.0 Neuromuscular Module scale was prepared in child self-report and parent report formats for children aged 5-18 years.The scale consists of a total of 25 items under 3 categories: symptoms related to neuromuscular disease, communication, and family resources.Items are scored on a Likert scale from 0 (never a problem) to 4 (always a problem).Higher scores on the module indicate better health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Ceyda Ulu, Principal Investigator — Gaziosmanpasa Research and Education Hospital
Locations (1):
- Gaziosmanpasa Research and Education Hospital, Istanbul, Gaziosmanpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yilmaz CU, Karabulut SS, Forestier FBE, Yalcinkaya EY. Effectiveness of aquatic therapy on balance and functionality in children with Duchenne and Becker muscular dystrophy : a prospective controlled pilot study. Dev Neurorehabil. 2026 Jan 31:1-8. doi: 10.1080/17518423.2026.2624412. Online ahead of print. PMID 41620441